CLINICAL TRIAL: NCT03867266
Title: Typical Atrial Flutter, Ablation Index and Point by Point Ablation
Acronym: FLAI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ospedale San Francesco (Other)
Responsible Party: Principal Investigator, Graziana Viola, Medical Doctor, Ospedale San Francesco
Other Study IDs: 73/2018
Record Dates: First submitted 2019-02-11; First posted 2019-03-07 (Actual); Last update posted 2019-03-07 (Actual); Status verified 2019-03

CONDITIONS: Typical Atrial Flutter
Keywords: Ablation index; Interlesion distance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Procedure: Ablation with radiofrequency — Ablation point by point on the cavo tricuspid isthmus guided by an index lesion

SUMMARY:
The Ablation of the typical atrial flutter can be considered substantially anatomical, the investigators want to test a protocol that foresees the use a lesion index (AI) and that respects the Inter-Lesion Distance (ILD) ≤ 6 mm on the cavo-tricuspid isthmus (CTI) The investigators want to prove how the introduction of a lesion index combined with the continuity of lesion can allow a "first pass block" of the CTI decreasing total Radio-Frequency (RF) times

DETAILED DESCRIPTION:
The Ablation of the typical atrial flutter can be considered substantially anatomical, the aim of the study is to test a protocol that foresees the use a lesion index and that respects the Inter-Lesion Distance ≤ 6 mm on the cavo-tricuspid isthmus to prove how the introduction of a lesion index combined with the continuity of lesion can allow a "first pass block" of the CTI decreasing total Radio-Frequency times With the aim of reducing the use of the fluoroscopy and ionizing radiations, an anatomical map of the right atrium will be reconstructed with a mapping catheter in all patients, and a 10-pole catheter will be placed in the coronary sinus.Then, the anatomy of the isthmus will be precisely defined with a catheter equipped with a force sensor ,identifying the tricuspid valve as the initial point of ablation and the inferior vena cava- right atrium junction as the end point of the line.Once the reconstruction has been completed, the ablation phase will start. Considering the values already validated for the left atrium, the protocol foresees the point-by-point ablation with the use of AI ≥ 500 and ILD≤ 6 mm.

The Visitag setting will be the following:

* Respiration Adjustment;
* Catheter Position Stability Min. Time = 3 sec, Max. Range = 5 mm;
* Force Over Time Time = 30% Min. Force = 4 gr. The power can be set between 35 and 40 watts. At the end of the isthmus ablation, line block will be evaluated by proximal CS pacing, acquiring at least 3 distinct points from the ablator catheter around the tricuspid annulus ,typically ostium of coronary sinus (CS), lateral tricuspid annulus and a point more proximal to the line of ablation.

Once this phase has been completed, 20 minutes of waiting time has to be considered. After this waiting time the block of the isthmus will be validated again with the same protocol described above.

Primary Endpoint -Anatomical first Pass block of the CTI.

Secondary Endpoint

-Reduction of procedural, RF and fluoroscopy times.

ELIGIBILITY:
Inclusion criteria:

* paroxysmal, persistent and /or long standing atrial flutter even in the presence of structural heart disease
* Informed consent form
* Age equal or above 18 years
* Skilled and willing to comply with all tests and follow up requirements
* Patients that ,in the context of ablation for fibrillation atrial, should also undergo to typical flutter ablation: in this case the data collected will be those related to typical flutter ablation.

Exclusion Criteria:

* Previous ablation for atrial flutter
* Atrial flutter secondary to electrolyte imbalance, thyroid disease or to a reversible or non-cardiac cause
* severe anemia,
* sepsis in progress
* Bypass procedure with coronary arterial artery in the last three months
* Pending cardiac transplantation or other cardiac surgery
* Pregnant or breastfeeding women
* Acute disease or active systemic infection or sepsis
* Documented left atrial thrombus
* Unstable angina
* Uncontrolled heart failure
* Life expectancy of less than 12 months
* Registration in any other study evaluating another device or medication
* Presence of intramural thrombi, tumor or other anomalies that preclude the introduction of the catheter into the vein system

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Caucasian population regardless gender
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2019-02-20 (Actual); Primary Completion 2019-06-01 (Estimated); Study Completion 2019-07-01 (Estimated)

PRIMARY OUTCOMES:
First pass block of the cavo tricuspid isthmus | 9 months
  Validation of the bidirectional block by pacing on the coronary sinus after completing the first line of the ablation

SECONDARY OUTCOMES:
radiofrequency time of application | 9 months
  reduction in radio frequency time in comparison with current literature
Near zero x ray | 9 months
  reduction of x-ray time
Procedural time | 9 months
  reduction in procedural time in comparison with current literature

CONTACTS AND LOCATIONS:
Locations (1):
- Ospedale San Francesco, Nuoro, Italy

IPD SHARING:
Plan to Share IPD: Undecided